CLINICAL TRIAL: NCT04728711
Title: A Double Masked, Placebo Controlled, Single Center, Randomized Clinical Trial to Assess the Safety and Efficacy of ADX-629 in Subjects With Mild Asthma Induced by the Bronchial Allergen Challenge (BAC)
Brief Title: A Double Masked, Placebo Controlled, Single Center, Randomized Clinical Trial to Assess the Safety and Efficacy of Subjects With Mild Asthma Induced by the Bronchial Allergen Challenge (BAC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-629-AA-001
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2023-01

CONDITIONS: Atopic Asthma
MeSH Terms: interventions — ADX-629

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ADX-629, 600 mg administered orally twice daily (PO bid) for a minimum of 1 week (Experimental)
  Interventions: Drug: ADX-629
- Placebo, 600 mg administered orally twice daily (PO bid) for minimum 1 week (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-629 — ADX-629, 600 mg administered orally twice daily (PO bid) for a minimum of 1 week
  Arms: ADX-629, 600 mg administered orally twice daily (PO bid) for a minimum of 1 week
Drug: Placebo — Placebo, 600 mg administered orally twice daily (PO bid) for minimum 1 week
  Arms: Placebo, 600 mg administered orally twice daily (PO bid) for minimum 1 week

SUMMARY:
A Double Masked, Placebo Controlled, Single Center, Randomized Clinical Trial to Assess the Safety and Efficacy of ADX-629 in Subjects with Mild Asthma Induced by the Bronchial Allergen Challenge (BAC)

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, between 18 to 65 years of age (inclusive) at Screening Visit.
* Subjects must give their signed and dated written informed consent (in English) to participate prior to commencing any study-related activities and must be willing to comply with study procedures, study restrictions, study protocol, and return for the required assessments.
* Female subjects of either non-childbearing potential or of child-bearing potential who commit to consistent and correct use of at least one highly effective or two effective forms of contraception starting at least 4 weeks prior to the Screening Visit and for at least 30 days post last dose of study drug.
* Generally healthy subjects with mild controlled asthma for 2 years at Screening Visit according to the Global Initiative for Asthma criteria.

Exclusion Criteria:

* History and presence of clinically significant cardiovascular, renal, neurologic, hepatologic, endocrinologic, gastrointestinal, genitourinary, autoimmune, hematological, or metabolic disease other than asthma, which in the opinion of Investigator may either put the subject at risk or influence the results during the study.
* Positive skin prick test to other perennial allergens (i.e., mold, dog with ≥ 3 mm wheal compared to negative control). Subjects with seasonal allergy symptoms that occur or are anticipated to occur during the study should result in subject exclusion or rescheduling until the subject is out of the allergy season.
* Any relevant pulmonary disease within 1 year prior to dosing at the discretion of the investigator.
* Recent hospitalization with asthma in the last 6 months or any other medical condition that the Investigator deems incompatible with participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight subjects were randomized in a crossover design trial.
Groups:
- First ADX-629, Then Placebo: ADX-629 300mg (milligrams) administered orally twice daily for one week, then a two-day washout, then placebo administered orally twice daily for one week.
- First Placebo, Then ADX-629: Placebo administered orally twice daily for one week, then a two-day washout, then ADX-629 300mg administered orally twice daily for one week.
Period: Overall Study
Arm/Group | First ADX-629, Then Placebo | First Placebo, Then ADX-629
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- First ADX-629, Then Placebo: ADX-629 300mg administered orally twice daily for one week, then a two-day washout, then placebo administered orally twice daily for one week.
- Total: Total of all reporting groups
Arm/Group | First ADX-629, Then Placebo | First Placebo, Then ADX-629 | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.0) | 34.0 (13.2) | 38.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.0 (4.9) | 30.33 (3.2) | 29.16 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: Safety was assessed through serious adverse event collection.
Time Frame: The safety assessment period was Day 1 - Day 7 for each treatment intervention.
Population: Safety population
Measure: Number; unit: participants
Groups:
- ADX-629: ADX-629 300mg administered orally twice daily for 1 week
- Placebo: Placebo administered orally twice daily for 1 week
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 8 | 8
participants | 0 | 0

2. Secondary Outcome: Change From Baseline in the Asthma Control Questionnaire
Description: Change from baseline in the asthma control questionnaire, which is seven questions on a seven-point scale (0 = totally controlled, 6 = extremely poorly controlled). The first six questions are answered by the subject. The seventh question, concerning forced expiratory volume in 1 second (FEV1) percentage predicted (0 = >95% predicted, 6 = <50% predicted), is completed by clinic staff. The asthma control questionnaire is calculated as the mean of the response to all seven questions, with a higher score being more severe.
Time Frame: The efficacy assessment period was Day 1 through Day 7 for each treatment period. Baseline is defined as the last non-missing assessment prior to randomization.
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale | -0.20 (0.41) | -0.05 (0.52)

3. Secondary Outcome: Change From Baseline in Sputum Eosinophils Percentage of Total Leukocytes
Description: Change from baseline in sputum eosinophils percentage of total leukocytes at seven hours post bronchial allergen challenge and 24 hours post bronchial allergen challenge. A reduction in sputum eosinophils percentage demonstrates improvement.
Time Frame: The efficacy assessment period was Day 1 through 7 for each treatment period. Baseline is defined as the last non-missing assessment prior to randomization.
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 8 | 8
percentage
  7 hours post-bronchial allergen challenge | 6.4 (8.8) | 11.6 (10.2)
  24 hours post-bronchial allergen challenge | 0.1 (1.8) | 16.2 (20.4)

4. Secondary Outcome: Change From Baseline in Sputum Neutrophils Percentage of Total Leukocytes
Description: Change from baseline in sputum neutrophils percentage of total leukocytes at 7 hours post bronchial allergen challenge and 24 hours post bronchial allergen challenge. A reduction in sputum neutrophils percentage demonstrates improvement.
Time Frame: as for outcome 2
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 8 | 8
percentage
  7 hours post-bronchial allergen challenge | -8.5 (16.1) | 4.3 (14.5)
  24 hours post-bronchial allergen challenge | 3.2 (18.6) | 7.8 (40.2)

ADVERSE EVENTS:
Time Frame: One week for each intervention
Groups:
- ADX-629: ADX-629 300 milligrams administered orally twice daily for 1 week
Arm/Group | ADX-629 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-629 (N=8) | Placebo (N=8)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT04728711/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT04728711/SAP_001.pdf